CLINICAL TRIAL: NCT04127526
Title: Connection to Environment With Cognitive Therapy (CONNECT): Exploring Trauma, Voices and Dissociation Through Targeted Psychological Intervention. A Single-Case Experimental Design
Brief Title: Psychological Therapy for Dissociation, Trauma and Voices: A Single Case Experimental Design
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN19MH346
Record Dates: First submitted 2019-10-04; First posted 2019-10-15 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Dissociation; Auditory Hallucination; Trauma, Psychological; Psychosis
Keywords: Dissociation; Psychosis; Trauma; Hallucinations; Psychological Therapies
MeSH Terms: conditions — Dissociative Disorders; Hallucinations; Psychological Trauma; Psychotic Disorders; Wounds and Injuries | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design. All participants will receive treatment and outcomes during treatment period will be compared to a randomized baseline period of two, three or four weeks (2 participant in each baseline arm).
Masking Description: Participants will be randomized to 3 baseline periods of two, three or four weeks. Both therapist (who is also the main researcher) and participant will be aware of which baseline arm the participant has been randomised to upon beginning the baseline, however not before this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Period of 2 weeks (Active Comparator): 2 participants will be randomly allocated to a baseline of 2 weeks before commencing CONNECT intervention.
  Interventions: Other: Connection to Environment with Cognitive Therapy (CONNECT)
- Baseline Period of 3 weeks (Active Comparator): 2 participants will be randomly allocated to a baseline of 3 weeks before commencing CONNECT intervention.
  Interventions: Other: Connection to Environment with Cognitive Therapy (CONNECT)
- Baseline Period of 4 weeks (Active Comparator): 2 participants will be randomly allocated to a baseline of 4 weeks before commencing CONNECT intervention.
  Interventions: Other: Connection to Environment with Cognitive Therapy (CONNECT)

INTERVENTIONS:
Other: Connection to Environment with Cognitive Therapy (CONNECT) — 8 sessions of strategies to reduce dissociation. Flexible, toolbox approach including but not limited to grounding strategies using objects, therapy oils and naming objects in the room.

SUMMARY:
Connection to Environment with Cognitive Therapy (CONNECT): A Single-Case Experimental Design Exploring Dissociative Experiences and Voices

Emerging empirical evidence has suggested that dissociation is a robust determinant of voice-hearing in psychosis, and that dissociation mediates the link between trauma and voices. Despite the emerging evidence-base, targeted therapeutic interventions focusing on dissociation remain largely untested.

The aim of the current study is to investigate whether targeting dissociation leads to improvements in distressing voices in people with a history of trauma. This will be done by delivering an eight session intervention called 'CONNECT' to six individuals within the Glasgow Psychological Trauma Service (GPTS) who hear voices, have experienced trauma and are dissociating. The intervention will focus on learning strategies to manage dissociation. It is hypothesised that reduced levels of dissociation will be associated with reduction in the frequency and distress associated with hearing voices.

This study will use a randomized multiple baseline single-case experimental design, meaning that participants will be randomly allocated to a baseline of two, three or four weeks and then will begin eight weeks of Connection to Environment Cognitive Therapy (CONNECT). As well as daily measures during baseline and intervention phases, there will be four assessment points (baseline, pre-intervention, post-intervention and follow-up). The study will take approximately three months plus follow-up one month after therapy ends. Individual levels of dissociation and voices will be compared during baseline and intervention periods using visual analysis and Tau-U.

This study will contribute to the evidence-based for dissociation interventions targeting distressing voices among this population. It serves to investigate the proposed mechanism in a clinical population using a therapeutic intervention. It will therefore inform clinicians of the effectiveness and feasibility of using such strategies in clinical practice and may have good generalizability to practice.

DETAILED DESCRIPTION:
1. Purpose and Design:

   We will use a single case experimental design (SCED). This approach is common in early stage studies when exploring whether an intervention creates therapeutic change, typically by applying multiple measures to investigate the constructs of interest. A SCED also offers advantages for this type of exploratory research over a randomized controlled trial (RCT), because of the rich detail in the data and reduced research costs. Also, because individuals are compared against their own baseline scores, a smaller sample can be recruited and participants do not need to be matched by age, education or other variables to have a comparable control group, like in a RCT. For a targeted intervention, like CONNECT, which is predicted to lead to change in voices, even after therapy has stopped, a multiple- baseline design is the most appropriate form of SCED. We will randomize participants to baseline periods of either two, three, or four weeks before the intervention begins. This increases confidence that any therapeutic change is more likely to be because of the intervention, not just natural change over time. Equally, if therapeutic change is demonstrated across participants allocated to different baseline lengths, we can be confident that it is not the length of the baseline that is responsible for this effect.

   Importantly, this study has been carefully designed in close partnership with the GPTS to ensure that it is in line with routine care. Open and close communication between the main researcher, the field supervisor and the wider team will be important to manage any ethical issues that may arise.
2. Aims and Hypotheses The aim of the current study is to investigate whether targeting dissociation through Connection to Environment Cognitive Therapy (CONNECT) is associated with improvements in distressing voices in people with a history of trauma. It is hypothesized that reductions in dissociation will lead to improvements in the frequency and distress associated with hearing voices.

   Primary Hypotheses:
   * Dissociation will significantly reduce following CONNECT therapy.
   * Voice frequency and distress will significantly reduce following CONNECT therapy.
   * Reductions in dissociation will precede reductions in voice frequency and distress

   Secondary Hypothesis:

   - CONNECT therapy will lead to increased perceived movement towards goals.
3. Plan of Investigation This study aims to investigate the above hypotheses by delivering a dissociation intervention to individuals who hear voices and have experienced trauma. The variables of interest will be monitored and compared within-participants between and within baseline and intervention phases. Follow-up data will be gathered one month after therapy. The intervention (CONNection to Environment with Cognitive Therapy:'CONNECT') was developed incorporating: a) interventions from current literature including previous work from a case-series of cognitive therapy in clients with trauma, dissociative experiences and distressing voices delivered in Manchester by Dr Varese and colleagues and b) interventions used in clinical practice in the GPTS. This information was gathered by means of a survey which was circulated by the researcher to the Glasgow Psychological Trauma Service (GPTS) staff in February 2019. The above information was collated to develop an integrated CONNECT manual that the therapist will utilize. CONNECT will adopt a 'toolbox' approach to learning strategies aimed to reduce dissociation and choice of strategies will therefore vary between participants, as this will be led by their individual preferences.

   Assessment and engagement (sessions 1-3) Early phases of intervention will focus on psych-education/normalization of voice-hearing and dissociative phenomena, and intervention strategies targeting dissociation

   Introducing strategies to target dissociative phenomena/processes (sessions 4-7) This phase of therapy emphasizes training and practice of skills to manage dissociative responses and increase perceived controllability of dissociation. This will be a 'toolbox' approach and therefore led by participant preference.

   Consolidation (session 8) This session directly follows intervention and focuses on consolidating prior learnings from intervention phase. This should consist of no additional learning of strategies to target dissociation. The purpose of this phase is to consider future care. Focus will therefore be on relapse prevention, risk management and linking in with other services or clinicians where appropriate.

   Review appointment There will also be a review appointment directly after CONNECT for the purpose of deciding future care. The field supervisor from the GPTS, Dr Kirsten Atherton, will be involved in this decision-making process and may also attend the appointment.

   Follow-up at 1 month There will be one appointment one month after CONNECT to re-administer measures and gain qualitative feedback of participation in therapy.
4. Recruitment:

   Potential participants will come into the study via and following their routine assessment pathway within the GPTS. The experimental intervention would be regarded as a 'phase 1 intervention' within the service. Individuals experiencing voices and dissociation would be offered the opportunity to participate in the study.

   If interested in taking part, the GPTS clinician will (with the individual's consent) pass on contact information to the main researcher, who will contact participants to arrange an information sharing appointment. Here, the study will be discussed in full with reference to the information sheet and any questions will be answered at this point. If interested in taking part, a follow-up consent appointment will be made whereby the participant will sign the consent form and fill in screening questionnaires to ascertain whether the person is suitable for the study based on the below inclusion/exclusion criteria.
5. Settings and Equipment:

   This study will be carried out during working hours in clinical rooms within the GPTS. Equipment will include participant information sheets, consent forms, paper copies of measures, paper, pens and a 'toolkit' consisting of various grounding objects e.g. aroma oils. A digital voice recorder belonging to the University of Glasgow will be used which is encrypted and password protected.
6. Procedure:

   This study utilises a randomized multiple baseline Single-Case Experimental Design (SCED) with assessment at four time points (baseline, start of intervention, end of intervention and follow-up). Randomisation: Participants will be randomised to baseline periods of two, three or four weeks using a pre-determined simple randomisation method. Randomisation will be completed using a computer-generated sequence before recruitment begins. The researcher will be blind to the baseline allocation until the point of consent and screening, when the researcher will open a sealed envelope to reveal this.

   All sessions will be audio recorded using an encrypted digital recorder provided by the University of Glasgow. Recordings will be used for supervision purposes to ensure the intervention is of high quality and to assess for content and fidelity of intervention.

   Interpreters will be accessed as part of routine practice within the GPTS. The researcher will endeavor to meet with the interpreter before the information sharing appointment to ensure minimal impact to the study procedure. The researcher will also endeavor for participants to have the same interpreter for the duration of the study. The field supervisor has noted this to be feasible within the GPTS.
7. Data Analysis:

   Tau-U analysis will be used to analyse changes in outcome variables between the four assessment time-points. Tau-U is a non-parametric rank order correlation statistic with promising application for SCED research. Visual data analyses will be conducted to analyse changes between and within phases. Visual analysis is routinely used in SCED research and will be conducted according to established guidelines.
8. Justification of Sample Size:

   This study aims to recruit a sample of six participants. As per SCED methodology, the participants in this study will serve as their own baseline. Guidelines for SCED research suggest that change ought to occur across a minimum of three participants, with a minimum of three time points per participant in order to account for between-participant variance and chance. Previous case series of a similar nature have included between nine and ten participants however participants in these studies did not have as much outcome data as the current study. Each participant in this study will have outcome data for four assessment points, as well as daily and in-session measures during baseline and intervention phases, thus having above the required three measures per phase. However, it is acknowledged that small sample size may result in limited generalizability to wider population. Therefore, demographic information will be taken into consideration when interpreting the results.
9. Ethical Issues:

   This study has undergone ethical review from the West of Scotland Research Ethical Committee (REC) and received approval (REC Reference: 19/WS/0125).
10. Dissemination:

The results will be submitted as part of the Doctorate in Clinical Psychology and will be read by staff from the Institute of Health and Wellbeing as well as external examiners. This work will be published in an academic journal, presented at conferences, and other clinical forums. As CONNECT is a new therapy, individual case reports may also be written and published in an academic journal to look at the feasibility and applicability of this therapy in more depth. Dissemination plans will be discussed with participants who will receive a summary of the results upon completion.

ELIGIBILITY:
Inclusion Criteria:

1. Voices: Hearing a voice/voices for a minimum of six months. Score ≥ 2 (i.e. "Voices occurring at least once a day") on the frequency item of the Psychotic Symptom Rating Scale (PSYRATS). Score ≥ 3 (i.e. "Voices are very distressing, although subject could feel worse") on the distress intensity rating of the PSYRATS.
2. Trauma: Score ≥ 1 on any of the items of the Brief Betrayal Trauma Survey-14 (BBTS-14) assessing lifetime exposure to interpersonal trauma.
3. Dissociation: Dissociative Experiences Scale Taxon (DES-T) score suggestive of clinical levels of dissociative symptoms, as indicated by a score > 20.
4. Treatment motivation: Indicated that they consider voices and dissociation as a presenting difficulty, and that they would like to receive a psychological intervention specifically designed to address these difficulties. This will be assessed using four items integrated in the PSYRATS interview administered and the self-reported therapy goals generated through the initial assessment in the GPTS.
5. Capacity to provide informed consent.
6. Deemed to have sufficient English to engage in therapy or have access to an appropriate interpreter within the GPTS.

Exclusion Criteria:

1. Concurrently receiving another form of psychological intervention.
2. Cognitive impairment that may impact ability to consent and/or engage.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Changes in Voices | Changes in voices measured from beginning to end of baseline; beginning to end of therapy and at 1 month follow-up
  Changes in voices will be measured using the Voice Hearing subscale of the Psychotic Symptom Rating Scale (PSYRATS; Haddock et al, 1999). This comprises of 12-items with responses ranging from 0 (absent) to 4 (severe).
Changes in Voices | Changes in voices measured in each session from beginning to end of baseline; beginning to end of therapy and at 1 month follow-up
  Voices will also be measured using a session measure as used in previous studies (Varese et al., 2012). This is a 5-item scale with questions on voice frequency, distress and control. Responses range from a scale of 0% to 100%.
Changes in Voices | Changes in voices measured daily from beginning to end of baseline and beginning to end of therapy
  Voices will also be measured using a daily self-report measure as used in previous studies (Varese et al., 2012). This consists of one question about voices "how much have the voices been a problem today?" with answers ranging from 0% (never) to 100% (always)
Changes in Dissociation | Changes in dissociation measured from beginning to end of baseline; beginning to end of therapy and at 1 month follow-up
  Changes in Dissociation will be measured using The Revised Dissociative Experiences Scale (DES-II, Carlson & Putnam, 1993). A 28-item, self-report measure of dissociative experiences in daily life with answers ranging from 0-100%.
Changes in Dissociation | Changes in dissociation measured in each session from beginning to end of baseline; beginning to end of therapy and at 1 month follow-up
  Changes in dissociation will also be measured using a session measure as used in previous studies (Varese et al., 2012). This includes seven questions relating to dissociative experiences in the past week, with answers ranging from 0% (never) to 100% (always).
Changes in Dissociation | Changes in dissociation measured daily from beginning to end of baseline and beginning to end of therapy
  Dissociation will also be measured using a daily self-report measure as used in previous studies (Varese et al., 2012). This consists of one question about dissociation "how much has dissociation been a problem today?" with answers ranging from 0% (never) to 100% (always).

SECONDARY OUTCOMES:
Changes in Psychological distress | Changes in distress measured from beginning to end of baseline; beginning to end of therapy and at 1 month follow-up
  Measured using the CORE-10 (Barkham et al, 2013). A 10-item scale of psychological distress, with four-point likert-responses. Will be administered at screening, beginning of baseline, beginning of therapy, end of therapy, 1 month follow-up
Changes in Therapeutic Alliance | Changes in Therapeutic Alliance measured from beginning to end of baseline; beginning to end of therapy and at 1 month follow-up
  Will be measured using the Working Alliance Inventory - Short Revised (Hatcher & Gillaspy, 2006). The WAI-SR is a self-report scale consisting of 12 items rated on a five-point likert scale. The WAI-SR has good reliability and validity with moderate correlation to clinical outcomes (r=0.24; Martin et al., 2000).
Changes in Perceived Movement Towards Goals | Changes in movement towards goals will be measured daily from beginning to end of baseline and beginning to end of therapy
  Changes in perceived movement towards personalized goals will be measured through the daily measure question "to what extent do you feel that you have moved towards your goal of X today?". Answers will range from 0% (not at all) to 100% (extremely)

OTHER OUTCOMES:
Participant experience: | This will be administered at 1-month follow up only
  Will be measured using Satisfaction with Therapy Questionnaire (STQ) (Lawlor et al., 2017). A 22-item self-report to assess satisfaction with CBTp. Items are scored on a scale ranging from 1 to 5, with higher scores corresponding to higher satisfaction
Trauma History | This will be administered at screening only
  Brief Betrayal Trauma Survey (BBTS; Goldberg & Freyd, 2006) is a 14-item self-report measure of frequency of traumatic experiences with responses ranging from 'never', 'one or two times' or 'more than that'.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gumley, Principal Investigator — University of Glasgow
Locations (1):
- NHS GG&C Glasgow Psychological Trauma Service (The Anchor), Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No